CLINICAL TRIAL: NCT07074132
Title: Impact of a Physical Activity Program on Body Composition, Strength, and Quality of Life in Postmenopausal Women
Brief Title: Physical Activity and Quality of Life in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wissal Abassi (Other)
Responsible Party: Sponsor-Investigator, Wissal Abassi, Principal Investigator, High Institute of Sports and Physical Education of Kef
Organization: High Institute of Sports and Physical Education of Kef (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PA-MenQL25
Record Dates: First submitted 2025-07-09; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-05

CONDITIONS: Quality of Life; Fitness Testing
Keywords: Obesity; Physical fitness; Long-term intervention; Combined exercise; Quality of life; Postmenopausal women
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): The experimental group performed a combined training program consisting of aerobic training at 50-70% of heart rate reserve (HRR) and muscle-strengthening training at 60-70% of one-repetition maximum (1-RM), three times per week for eight months.
  Interventions: Behavioral: Combined Aerobic and Muscle-Strengthening Training Program
- Control group (No Intervention): No training intervention was intended for the control group.

INTERVENTIONS:
Behavioral: Combined Aerobic and Muscle-Strengthening Training Program — A combined training program including both aerobic and muscle-strengthening physical activities within the same session, conducted over a period of 8 months. Aerobic training is performed at an intensity of 50-70% of heart rate reserve (HRR), and strength training at 60-70% of one-repetition maximum (1-RM). The training is conducted three times per week.
  Arms: Training group

SUMMARY:
The goal of this clinical trial is to investigate the effects of a combined aerobic and muscle-strengthening training program on body composition, physical fitness, and quality of life in overweight or obese postmenopausal women. The main question it aims to answer is: Does this training modality improve body composition, enhance physical fitness, and increase quality of life in this population ? Researchers will compare outcomes between an experimental group following the training protocol and a control group with no training intervention, in order to determine whether the program leads to measurable improvements in these parameters. Participants in the training group will engage in aerobic exercise at 50-70% of heart rate reserve (HRR) and strength training at 60-70% of one-repetition maximum (1-RM), three times per week for 8 months.

Participants in the control group will not engage in any structured physical training and will be asked to maintain their usual daily routines.

DETAILED DESCRIPTION:
Overweight and obesity in postmenopausal women are associated with adverse changes in body composition, decreased physical fitness, and a decline in overall quality of life. The postmenopausal period is marked by hormonal changes that contribute to increased fat accumulation, loss of muscle mass, and heightened vulnerability to metabolic and cardiovascular diseases. These changes often lead to reduced functional capacity and well-being. Although exercise has been widely recognized as an effective strategy for improving health outcomes, there is a lack of long-term intervention studies combining aerobic and strength training in this specific population. The purpose of this clinical trial is to investigate the effects of a combined aerobic and muscle-strengthening training program for 8 months on body composition, physical fitness, and quality of life in overweight or obese postmenopausal women.

Thirty-six overweight/obese postmenopausal women were randomly assigned to either a training (n = 18), or a control group (n = 18). The training group will engage in aerobic exercise at 50-70% HRR and strength training at 60-70% 1-RM, three times per week for eight months. The control group will not participate in any structured physical training and will be instructed to maintain their usual lifestyle habits. Assessments of body composition, physical fitness, and quality of life were assessed before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age range (50-62 years).
* Postmenopausal women (absence of menstruation > 12 months).
* Body mass index (BMI) ≥ 25 kg/m².
* Body weight remained constant (±2 kg) for the past 3 months.
* Stable dietary habits and physical activity for at least 3 months.
* Sedentary lifestyle (physical activity less than 1 hour per week).

Exclusion Criteria:

* Medical contraindications to physical activity.
* Metabolic, hormonal, orthopedic, or cardiovascular diseases.
* Current use of hormone replacement therapy or any prescribed medication.

Ages: 50 Years to 62 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 36 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Body weight | Baseline (Day 0) and after 8 months of intervention.
  Body weight (kg) was recorded with participants barefoot and wearing light clothing, using the InBody 270 bioelectrical impedance device (InBody, Cerritos, CA, USA).
Body fat | Baseline (Day 0) and after 8 months of intervention.
  Body fat (%) was recorded using the InBody 270 bioelectrical impedance device (InBody, Cerritos, CA, USA).
Body mass index | Baseline (Day 0) and after 8 months of intervention.
  Body mass index (kg/m²) was calculated as weight (kg) divided by height squared (m²).
Lean mass | Baseline (Day 0) and after 8 months of intervention.
  Lean mass (%) was recorded with participants barefoot and wearing light clothing, using the InBody 270 bioelectrical impedance device (InBody, Cerritos, CA, USA).
Basal metabolic rate | Baseline (Day 0) and after 8 months of intervention.
  Basal metabolic rate (kcal/day) was assessed using the InBody 270 bioelectrical impedance device (InBody, Cerritos, CA, USA).
Aerobic Capacity | Baseline (Day 0) and after 8 months of intervention.
  Aerobic capacity was assessed using the 6-minute walk test (6MWT), administered according to standardized procedures, with participants walking on a flat, straight course for six minutes.
Lower limb functional strength. | Baseline (Day 0) and after 8 months of intervention.
  Lower limb functional strength was assessed using the 30-Second Chair Stand Test.
Agility and dynamic balance | Baseline (Day 0) and after 8 months of intervention.
  Agility and dynamic balance were assessed using the 8-Foot Up and Go (8UG) test.
Quality of life (SF-36 Questionnaire) | Baseline (Day 0) and after 8 months of intervention.
  Quality of life was assessed using the Short Form Health Survey 36 (SF-36), a validated 36-item questionnaire measuring physical and mental health domains.

CONTACTS AND LOCATIONS:
Overall Officials: Antonella MUSCELLA, Professor, Principal Investigator — Department of Biological and Environmental Science and Technologies (DiSTeBA), University of Salento, 73100 Lecce, Italy.; Wissal Abassi, Dr, Principal Investigator — Research Unit "Sport Sciences, Health and Movement"(UR22JS01) High Institute of Sport and Physical Education of Kef, University of Jendouba, 7100 Kef, Tunisia.
Locations (1):
- Department of Biological and Environmental Sciences and Technologies (DiSTeBA), University of Salento, Centro Ecotekne, Pal. B S.P. 6, Lecce, LE (Lecce), Italy

IPD SHARING:
Plan to Share IPD: No
For confidentiality reasons, all data from this study are available upon request.